CLINICAL TRIAL: NCT05255835
Title: A Randomized Prospective Study to Evaluate the Effect of Semiconductor Knee Sleeves on Pain in Osteoarthritis of the Knee.
Brief Title: The Effect of Semiconductor Knee Sleeves on Pain in Osteoarthritis of the Knee.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Mikkel Rathsach Andersen, MD., Ph.D., Associate prof., Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-20080028
Record Dates: First submitted 2022-01-06; First posted 2022-02-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee
Keywords: Knee; Arthrosis; Pain; Osteoarthritis; Knee-Sleeves; Semiconductor
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Investigated knee sleeves appear identical, a printed code reveals to investigator if knee sleeves contains semiconductors (intervention group) or are cotton only (placebo group).
  Participants, care provider and outcome assessors are blinded to intervention/placebo grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semiconductor knee-sleeves (Active Comparator): Knee-sleeves containing semiconductor elements within the fabric constitute the intervention arm.
  Interventions: Device: Semiconductor Knee Sleeves
- Placebo knee-sleeves (Placebo Comparator): Cotton knee-sleeves constitute the placebo arm.
  Interventions: Device: Cotton Knee Sleeves (Placebo)

INTERVENTIONS:
Device: Semiconductor Knee Sleeves — semiconductor elements germanium and carbon within the cotton fabric
  Other Names: Incrediwear
  Arms: Semiconductor knee-sleeves
Device: Cotton Knee Sleeves (Placebo) — cotton fabric knee sleeves
  Other Names: Incrediwear (Placebo)
  Arms: Placebo knee-sleeves

SUMMARY:
To assess the benefits of using semiconductor (germanium and carbon) woven knee sleeves products in patients with osteoarthritis of the knee. To compare patients in a blinded randomized trial with and without the semiconductor knee sleeves product during the first 3 months period after initial contact at the outpatient clinic.

Aims:

The hypothesis of the study is that the semiconductor sleeve will reduce pain and improve knee function in active group when compared to the placebo group.

DETAILED DESCRIPTION:
Semiconductor woven knee sleeves work by increasing circulation to reduce inflammation, relieve pain, optimize performance, and accelerate recovery. Unlike compression products, semiconductor knee sleeves do not need to compress to work. Instead, the technology incorporates the semiconductor elements germanium and carbon within the fabric, which when stimulated by body heat, by release of negative ions. The negative ions activate molecular vibrations that increase blood flow and speed. Increasing circulation helps bring more oxygen and nutrients to the target area, which optimizes the body's natural healing process and accelerates recovery. Benefits of Increased Blood Circulation Include:

* Accelerated Recovery
* Reduced Swelling
* Optimized Performance
* Reduced Fatigue
* Thermoregulation

Investigators wish to investigate a possible effect on knee pain and function in patients with osteoarthritis of the knee.

Subject Enrollment:

Subjects referred with arthrosis of the knee to the out-patient clinic, at the Hip- and Knee-arthroplasty Unit, Herlev Gentofte Hospital. Included subjects must be assessed by an arthroplasty surgeon to have arthrosis without present indication for surgery, and to be eligible for a period of conservative treatment including physiotherapist guided training and paracetamol treatment.

This is a prospective study that will require informed consent.

Study size calculation A 25% difference in pain reduction between the intervention group compared and the placebo group is considered clinically relevant. Standard deviation expected at 25 mm on a 100 mm visual analog scale (VAS) for pain1. A type II error set at 10%, and a two-sided 5% significance level. A total number of 36 subjects with 18 in each group was calculated. To account for dropouts and the risk of conversion to surgical strategy during the follow-up period we plan to enroll a total of 25 subjects in each group.

Study Population: Estimated enrollment Target enrollment - 50 patients

* 25 patients with the semiconductor knee sleeve.
* 25 patients with the placebo sleeve.

ELIGIBILITY:
Inclusion Criteria:

* Arthrosis of the Knee
* Surgery not yet indicated
* 40-90 years old
* Male or female
* Compliant patient
* BMI less than 35
* Able to understand Danish sufficiently for written consent

Exclusion Criteria:

* Rheumatoid Arthritis
* Previous blood clots
* BMI greater than 35
* Varicosities on operative leg

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Knee Pain | 3 months
  Visual Analog Scale 0-100, 0-no pain, 100 maximum pain

SECONDARY OUTCOMES:
Knee function | 3 months
  Oxford Knee Score, 0-48, 0-indication of low level of knee function, 48 indication of satisfactory knee function
Knee Range of Motion (ROM) | 3 months
  Range of motion for the knee, extension-flexion- 0-140
Life Quality assessment | 3 months
  SF-36 score, (Short Form Survey-36), 36 life quality items questionaire, 0-lowest score, 100-highest score

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel R Andersen, MD., Ph.D., Study Chair — Gentofte Hospital; Mathias R Vergmann, Physiotherapeut, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
All study results will be published